CLINICAL TRIAL: NCT00933686
Title: Growth Hormone Treatment of Severe Fibromyalgia Syndrome Associated With Functional Failure of Somatotropic Axis. A Multicentre, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Growth Hormone in Neuroendocrine Dysfunction With Severe Fibromyalgia Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck, S.L., Spain (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 27560
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Saizen® (Active Comparator)
  Interventions: Drug: Saizen®
- Placebo + Saizen® (Active Comparator)
  Interventions: Drug: Placebo and Saizen®

INTERVENTIONS:
Drug: Saizen® — Saizen® (Somatropin) 0.006 milligram per kilogram (mg/kg) will be administered subcutaneously daily for 12 months. Dose will be titrated (an increase of 0.2 milligram per day) if the increase in insulin-like growth factor 1 (IGF-1) is less than 50 percent of the baseline value. Dose titrations will be made at Month 1, 3, 7 and 9.
  Other Names: Somatropin
  Arms: Saizen®
Drug: Placebo and Saizen® — Placebo matched to Saizen® will be administered for the first 6 months followed by treatment with Saizen® (Somatropin) 0.006 mg/kg subcutaneously daily for next 6 months. Saizen® dose will be titrated (an increase of 0.2 milligram per day) if the increase in insulin-like growth factor 1 (IGF-1) is less than 50 percent of the baseline value. Dose titrations will be made at Month 7 and 9.
  Arms: Placebo + Saizen®

SUMMARY:
The purpose of this study is to evaluate the efficacy of recombinant human growth hormone (r-hGH) treatment in severe fibromyalgia subjects with growth axis dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Women aged greater than or equal (>=) 18 years
* Fibromyalgia diagnosed at least one year before
* History of generalized pain and at least 16 positive tender points (1990 American College of Rheumatology [ACR] criteria)
* Body Mass Index (BMI) less than or equal to(=<) 32
* Normal GH stimulation test (insulin)
* Stable (>= 3 months unchanged) standard treatment with amitriptyline (10-50 milligram per day [mg/day]) plus selective serotonin reuptake inhibitor (10-40 mg/day) plus tramadol (25-400 mg/day)
* Active rehabilitation program during the previous year (at least 30 minutes/day)
* Fibromyalgia Impact Questionnaire (FIQ) score >=75
* IGF-1 serum level =< 150 nanogram/milliliter (ng/mL) otherwise =< 2 SD of the local lab normality)
* Normal response to IGF-1 generation test
* Chronic Fatigue Symptoms (Multidimensional Assessment of Fatigue [MAF])
* Effective anti-conception
* Willingness to comply with the protocol
* Written Informed consent

Exclusion Criteria:

* Major psychiatric condition
* Rheumatic disease, including systemic lupus erythematosus (SLE)
* Previous or current malignancies, active or inactive
* Clinical history intracranial space occupying lesion
* Reactive or secondary (rheumatoid arthritis [RA], osteoarthritis) fibromyalgia syndrome (FMS)
* Antinuclear antibody (ANA) greater than or equal 1:80
* Abnormal Creatine phosphokinase (CPK) or aldolase serum levels
* Not controlled thyroid disease in the last 3 months (free Thyroxine [T4] and Thyrotrophin-stimulating hormone [TSH] serum levels)
* Diabetes mellitus
* Adrenal gland disease (any abnormal cortisolemia, will be confirmed by 24-hour cortisoluria)
* Pregnancy or breast feeding
* Known to be hypersensitive to somatotropin or any of the excipients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2007-12; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillem Cuatrecasas, MD, Principal Investigator — Centro Medico Teknon
Locations (1):
- Centro Medico Teknon, Endocrinology Department, Barcelona, Spain

REFERENCES:
- [Derived] Cuatrecasas G, Alegre C, Fernandez-Sola J, Gonzalez MJ, Garcia-Fructuoso F, Poca-Dias V, Nadal A, Cuatrecasas G, Navarro F, Mera A, Lage M, Peino R, Casanueva F, Linan C, Sesmilo G, Coves MJ, Izquierdo JP, Alvarez I, Granados E, Puig-Domingo M. Growth hormone treatment for sustained pain reduction and improvement in quality of life in severe fibromyalgia. Pain. 2012 Jul;153(7):1382-1389. doi: 10.1016/j.pain.2012.02.012. Epub 2012 Mar 31. PMID 22465047
- [Derived] Cuatrecasas G, Gonzalez MJ, Alegre C, Sesmilo G, Fernandez-Sola J, Casanueva FF, Garcia-Fructuoso F, Poca-Dias V, Izquierdo JP, Puig-Domingo M. High prevalence of growth hormone deficiency in severe fibromyalgia syndromes. J Clin Endocrinol Metab. 2010 Sep;95(9):4331-7. doi: 10.1210/jc.2010-0061. Epub 2010 Jul 14. PMID 20631018

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 subjects were enrolled of whom 113 subjects were randomised and treated.
Groups:
- Saizen®: Saizen® (Somatropin) 0.006 milligram per kilogram (mg/kg) was administered subcutaneously daily for 12 months. Saizen® dose was titrated (an increase of 0.2 milligram per day) if the increase in insulin-like growth factor 1 (IGF-1) was less than 50 percent of the baseline value. Dose titrations were made at Month 1, 3, 7 and 9.
- Placebo + Saizen®: Placebo matched to Saizen® was administered for the first 6 months followed by treatment with Saizen® (Somatropin) 0.006 mg/kg subcutaneously daily for next 6 months. Saizen® dose was titrated (an increase of 0.2 milligram per day) if the increase in IGF-1 was less than 50 percent of the baseline value. Dose titrations were made at Month 7 and 9.
Period: Overall Study
Arm/Group | Saizen® | Placebo + Saizen®
Started | 55 | 58
Completed | 45 | 47
Not Completed | 10 | 11
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Failure to show up at endpoint visits | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saizen® | Placebo + Saizen® | Total
Number analyzed (Participants) | 55 | 58 | 113
Age Continuous [Mean (Standard Deviation); unit: years] | 49.9 (9.5) | 50.3 (9.6) | 50.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Less Than 11 Tender Points at Month 6
Description: The musculoskeletal component in form of pain on palpation in at least 11 of 18 tender point sites is required to fulfill the American College of Rheumatology (ACR) criteria for fibromyalgia syndrome, An important response is considered when the number of tender points falls below 11 since it is the threshold for fibromyalgia diagnosis.
Time Frame: Month 6
Population: Intention-to-treat (ITT) population included all the participants who were randomized in the study. 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 51 | 50
Percentage of participants | 20 | 22

2. Primary Outcome: Percentage of Participants With Less Than 11 Tender Points at Month 12
Description: The musculoskeletal component in form of pain on palpation in at least 11 of 18 tender point sites is required to fulfill the ACR criteria for fibromyalgia syndrome, An important response is considered when the number of tender points falls below 11 since it is the threshold for fibromyalgia diagnosis.
Time Frame: Month 12
Population: ITT population included all the participants who were randomized in the study. 'N' signifies number of participants who were evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 45 | 47
Percentage of participants | 53 | 34

3. Secondary Outcome: Fibromyalgia Impact Questionnaire (FIQ) Total Score
Description: Fibromyalgia Impact Questionnaire (FIQ) is a 10-item questionnaire that measures physical impairment, well-being, missed work, pain, fatigue, rest, stiffness, anxiety, and depression. Score ranges from 0 (best result - very well) to 100 (worst result - awful).
Time Frame: Baseline, Month 1, 3, 6, 7, 9 and 12
Population: ITT population included all the participants who were randomized in the study. 'N' signifies number of participants who were evaluable for this outcome measure. 'n' signifies number of participants who were evaluable at each time-point for each arm group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 54 | 57
Units on a scale
  Baseline (n=54, 57) | 85.7 (2.3) | 86.0 (1.8)
  Month 1 (n=52, 54) | 74.6 (3.6) | 73.3 (4.7)
  Month 3 (n=52, 54) | 72.1 (4.4) | 66.4 (5.1)
  Month 6 (n=51, 50) | 65.8 (4.8) | 68.4 (5.3)
  Month 7 (n=51, 50) | 59.2 (5.5) | 65.8 (5.7)
  Month 9 (n=51, 50) | 58.2 (6.4) | 65.1 (5.7)
  Month 12 (n=45, 47) | 52.5 (6.5) | 64.7 (6.5)

4. Secondary Outcome: Visual Analog Scale (VAS) Total Score
Description: Visual Analog Scale (VAS) is a 100 millimeter (mm) scale. Intensity of pain range: 0 mm=no pain to 100 mm=worst possible pain.
Time Frame: Baseline, Month 1, 3, 6, 7, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 54 | 57
mm
  Baseline (n=54, 57) | 73.3 (3.4) | 74.3 (3.1)
  Month 1 (n=52, 54) | 65.1 (4.2) | 68.0 (5.7)
  Month 3 (n=52, 54) | 63.7 (5.6) | 58.4 (5.8)
  Month 6 (n=51, 50) | 57.6 (5.7) | 60.4 (6.6)
  Month 7 (n=51, 50) | 54.6 (5.2) | 56.1 (6.2)
  Month 9 (n=51, 50) | 51.2 (6.7) | 60.3 (6.3)
  Month 12 (n=45, 47) | 45.0 (6.9) | 60.6 (6.0)

5. Secondary Outcome: EuroQol 5-Dimensions (EQ-5D) Total Score
Description: EuroQol 5-Dimensions (EQ-5D) questionnaire is a measure of health status and quality of life (QoL). The EQ-5D defines health in terms of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Score range for each item is 0 to 3, with 3 being the most severe. Total score range is 0 to 15. Lower scores represent a better QoL.
Time Frame: Baseline, Month 1, 3, 6, 7, 9 and 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 54 | 57
Units on a scale
  Baseline (n=54, 57) | 11.07 (0.44) | 11.24 (0.42)
  Month 1 (n=52, 54) | 10.46 (0.45) | 10.45 (0.42)
  Month 3 (n=52, 54) | 10.13 (0.45) | 10.06 (0.55)
  Month 6 (n=51, 50) | 10.00 (0.48) | 10.16 (0.56)
  Month 7 (n=51, 50) | 9.63 (0.49) | 9.77 (0.54)
  Month 9 (n=51, 50) | 9.49 (0.60) | 9.80 (0.50)
  Month 12 (n=45, 47) | 9.09 (0.64) | 9.94 (0.56)

6. Secondary Outcome: Multidimensional Assessment of Fatigue (MAF) Total Score
Description: Multidimensional Assessment of Fatigue (MAF) consists of 16 questions. The score range for first 14 questions is between 0 and 10 for each question while for the last two questions it is 0 and 4 for each question. Total score range for first 14 questions is 0 to 100 and for last two questions is 0 to 8. Lower scores on the each represent the better participant's condition, whereas, higher scores indicate worsening condition.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 3
Measure: Number; unit: Units on a scale
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 54 | 57
Units on a scale
  1 to 14 questions: Baseline (n=54, 57) | 90 | 83
  1 to 14 questions: Month 6 (n=51, 50) | 85 | 78
  1 to 14 questions: Month 12 (n=45, 47) | 73 | 78
  15 and 16 question: Baseline (n=54, 57) | 7 | 7
  15 and 16 question: Month 6 (n=51, 50) | 6 | 6
  15 and 16 question: Month 12 (n=45, 47) | 5 | 6

7. Secondary Outcome: Percentage of Participants With Positive Response on Quality of Life Assessment of Growth Hormone [GH] Deficiency in Adults (QoL AGHDA) Scale
Description: Quality of Life Assessment of GH Deficiency in Adults (QoL AGHDA) questionnaire consists of 25 items that evoke yes or no answers. A score of 1 is given to each item affirmed and these are summed to give the total score. The maximum score is 25, which represents a poor quality of life. The minimum score is 0, which represents a good quality of life. Each question has to be answered with a NO/YES and for each YES, one point is added. The more YES, the higher the score and the worse. Decrease in the positive responses is an index of improvement. So, when the percentage of positive responses on the scale decreases, it is considered a response rate.
Time Frame: Baseline, Month 6 and 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Saizen® | Placebo + Saizen®
Number analyzed (Participants) | 54 | 57
Percentage of participants
  Baseline (n=54, 57) | 73 | 72
  Month 6 (n=51, 50) | 70 | 69
  Month 12 (n=45, 47) | 59 | 70

ADVERSE EVENTS:
Time Frame: Baseline up to Month 12
Arm/Group | Saizen® | Placebo + Saizen®
Serious Adverse Events (participants affected / at risk) | 4/55 | 0/58
Other Adverse Events (participants affected / at risk) | 45/55 | 51/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=55) | Placebo + Saizen® (N=58)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sleep apnoea syndrome (Nervous system disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Food allergy (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saizen® (N=55) | Placebo + Saizen® (N=58)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 8
Otitis media acute (Ear and labyrinth disorders) | 1 | 0
Dizziness (Ear and labyrinth disorders) | 0 | 5
Ear infection (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Aptyalism (Gastrointestinal disorders) | 1 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 7
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 2
Dysgeusia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Acetonaemic vomiting (Gastrointestinal disorders) | 0 | 2
Pain exacerbated (General disorders) | 5 | 5
Pain (General disorders) | 2 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 5
Fall (General disorders) | 0 | 2
Malaise (General disorders) | 0 | 1
Transaminases increased (Hepatobiliary disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Vaginal candidiasis (Infections and infestations) | 4 | 0
Gastroenteritis (Infections and infestations) | 0 | 3
Corneal infection (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 0 | 1
Injury asphyxiation (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthroscopy (Investigations) | 1 | 0
Blood pressure systolic increased (Investigations) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 8
Oedema (Musculoskeletal and connective tissue disorders) | 17 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Trigger finger (Musculoskeletal and connective tissue disorders) | 3 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 16
Humerus fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pelvic fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Radius fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 5
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Epicondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ganglion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle rupture (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Wrist deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polyp colorectal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 21 | 13
Paraesthesia (Nervous system disorders) | 13 | 6
Insomnia (Nervous system disorders) | 9 | 2
Carpal tunnel syndrome (Nervous system disorders) | 8 | 7
Somnolence (Nervous system disorders) | 2 | 4
Sciatica (Nervous system disorders) | 2 | 0
Syncope (Nervous system disorders) | 0 | 6
Migraine (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 0 | 2
Dysphemia (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 5 | 0
Amnesia (Psychiatric disorders) | 3 | 0
Depression (Psychiatric disorders) | 2 | 1
Sleep talking (Psychiatric disorders) | 1 | 0
Memory impairment (Psychiatric disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 7 | 1
Cystitis (Renal and urinary disorders) | 3 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 2 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 4
Hypertrophy breast (Reproductive system and breast disorders) | 0 | 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Furuncle (Skin and subcutaneous tissue disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Impaired work ability (Social circumstances) | 5 | 7
Wheelchair user (Social circumstances) | 0 | 1
Hypertension (Vascular disorders) | 4 | 1
Hot flush (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other